CLINICAL TRIAL: NCT06864026
Title: A Phase 4, Prospective, Open-Label, Single-Arm Study to Assess the Effectiveness of Tirzepatide After Initiation of Ixekizumab in Adult Participants With Active Psoriatic Arthritis and Overweight or Obesity in Clinical Practice.
Brief Title: A Study to Investigate Effectiveness of Tirzepatide Following Initiation of Ixekizumab in Participants With Active Psoriatic Arthritis and Overweight or Obesity in Clinical Practice (TOGETHER AMPLIFY-PsA)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27350; I1F-MC-RHDE (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Psoriatic Arthritis; Overweight or Obesity
MeSH Terms: conditions — Arthritis, Psoriatic; Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirzepatide (Experimental): Participants will continue on ixekizumab and take tirzepatide administered subcutaneously (SC) as per label.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176

SUMMARY:
The main purpose of this study is to assess the effectiveness of adding tirzepatide to ixekizumab therapy in standard clinical practice in participants with moderate-to-severe PsA and obesity or overweight with at least 1 weight-related comorbidity.

The study will last up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of active psoriatic arthritis (PsA) as defined by a rheumatologist or other healthcare professional (HCP) experienced in treating PsA.
* Body Mass Index (BMI) of 30 kilograms per meter squared (kg/m²) or greater (obesity) or 27 kg/m2 to <30 kg/m² (overweight) in the presence of at least 1 weight-related comorbid condition (hypertension, dyslipidemia, type 2 diabetes, obstructive sleep apnea, or cardiovascular disease).
* Who have been treated with ixekizumab for approximately 3 months (±1 month) prior to decision to add tirzepatide.
* Must be able to initiate tirzepatide (Day 0) within 30 days of treatment decision (baseline or screening).

Exclusion Criteria:

* Have currently received ixekizumab for more than 4 months or less than 2 months.
* Had any exposure to tirzepatide or other glucagon-like peptide-1 (GLP-1) receptor agonist (for example, dulaglutide, liraglutide, or semaglutide).
* Are currently enrolled in any other clinical study.
* Have a known hypersensitivity to any component of tirzepatide.
* Have a personal or family history of medullary thyroid cancer.
* Have multiple endocrine neoplasia type 2.
* Have type 1 diabetes mellitus.
* Have a history of chronic or acute pancreatitis at any time before screening.
* Have a history of proliferative diabetic retinopathy, diabetic maculopathy, or nonproliferative diabetic retinopathy that requires acute treatment.
* Have a history of ketoacidosis or hyperosmolar state/coma.
* Have a history of severe hypoglycemia unawareness within the 6 months before screening.
* Have a history of severe gastrointestinal complications, including gastroparesis, gastroesophageal reflux disease, dyspepsia, chronic nausea/vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Normalized Functioning Health Assessment Questionnaire - Disability Index (HAQ-DI) ≤0.5 at 12 Months of Therapy | 12 Months
  The HAQ-DI is a patient-reported outcome questionnaire that is used to measure disease associated disability as an assessment of physical function. It consists of 20 questions referring to 8 domains of functioning. Participants assess their degree of difficulty when performing the activities over the past week on a 4-item ordinal scale, ranging from 0, "without any difficulty," to 3, "unable to do." The scores of each of the 8 domains are summed and divided by 8. Higher scores indicate more limitations in physical function.
Percentage of Participants Achieving at Least a 10% Weight Loss at 12 Months of Therapy | 12 Months
  Percentage of participants achieving at least a 10% weight loss at 12 months of therapy.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Tender Joint Count (TJC) ≤1 | Month 6 and Month 12
  Percentage of participants achieving TJC ≤1.
Percentage of Participants Achieving Swollen Joint Count (SJC) ≤1 | Month 6 and Month 12
  Percentage of participants achieving SJC ≤1.
Percentage of Participants Achieving Body Surface Area (BSA) ≤3% | Month 6 and Month 12
  Percentage of participants achieving BSA ≤3%.
Percentage of Participants Achieving Patient Global Assessment of Disease Activity Numeric Rating Score (PaGADA NRS) of ≤2 | Month 6 and Month 12
  The PaGADA NRS is an 11-point scale from 0 to 10 that is anchored by 2 verbal descriptors, "very well" and "very poor." Higher scores represent a higher level of disease activity.
Percentage of Participants Achieving Patient Pain Visual Analogue Scale (VAS) ≤15 | Month 6 and Month 12
  The Patient's Assessment of Arthritis Pain is a single-item, patient-reported outcome instrument, used to access the current severity of participants' joint pain in relation to their PsA on a horizontal VAS of 0 to 100 mm. The Patient's Assessment of Arthritis Pain is anchored by 2 verbal descriptors, "no pain" and "as severe as can imagine."
Percentage of Participants Achieving Physician Global Assessment of Disease Activity (PhGADA) NRS ≤2 | Month 6 and Month 12
  The PhGADA NRS is an 11-point scale anchored by 2 verbal descriptors, "none" and "extremely active disease."
Percentage of Participants Achieving HAQ-DI Sore ≤0.5 and at Least a 10% Weight Loss | Month 6 and Month 12
  The HAQ-DI is a patient-reported outcome questionnaire that is used to measure disease associated disability as an assessment of physical function. It consists of 20 questions referring to 8 domains of functioning. Participants assess their degree of difficulty when performing the activities over the past week on a 4-item ordinal scale, ranging from 0, "without any difficulty," to 3, "unable to do." The scores of each of the 8 domains are summed and divided by 8. Higher scores indicate more limitations in physical function.
Percentage of Participants With a Functional Assessment of Chronic Illness Therapy (FACIT) -Fatigue With ≥4-point Increase from Baseline | Month 6 and Month 12
  FACIT-F is a patient-reported, 13-item questionnaire that specifically assess the self-reported severity of fatigue and its impact upon daily activities and functioning. The FACIT-F uses 0 ("not at all") to 4 ("very much") Likert scale to assess fatigue and its impact in the past 7 days. Total score ranges from 0 to 52, based on a rating of 5-point Likert scale. Scores for negatively worded items are reversed, such that higher scores are better (that is, less fatigue).
Percentage of Participants With a Short-Form 36 (SF36) Physical Component Score (PCS) Minimum Clinically Important Difference (MCID) | Month 6 and Month 12
  The SF-36v2 acute form is a 36-item, generic, patient-completed measure designed to assess health-related quality of life with 8 health domains. Items are rated on 3-, 5-, or 6-point Likert scales. Each domain is individually scored by summing item responses and transforming them to a 0-100 scale. The eight domains are aggregated into two summary scores: Physical and Mental Component Summaries. Each summary score is norm based and presented in the form of T-scores, with a mean of 50 and a standard deviation of 10, with higher scores indicating better health status or functioning.
Percentage of Participants With a Short-Form 36 (SF36) Mental Component Score (MCS) MCID | Month 6 and Month 12
  The SF-36v2 acute form is a 36-item, generic, patient-completed measure designed to assess health-related quality of life with 8 health domains. Items are rated on 3-, 5-, or 6-point Likert scales. Each domain is individually scored by summing item responses and transforming them to a 0-100 scale. The eight domains are aggregated into two summary scores: Physical and Mental Component Summaries. Each summary score is norm based and presented in the form of T-scores, with a mean of 50 and a standard deviation of 10, with higher scores indicating better health status or functioning.
Percentage of Participants Achieving a HAQ-DI score ≤0.5 | Month 6
  The HAQ-DI is a patient-reported outcome questionnaire that is used to measure disease associated disability as an assessment of physical function. It consists of 20 questions referring to 8 domains of functioning. Participants assess their degree of difficulty when performing the activities over the past week on a 4-item ordinal scale, ranging from 0, "without any difficulty," to 3, "unable to do." The scores of each of the 8 domains are summed and divided by 8. Higher scores indicate more limitations in physical function.
Percentage of Participants with ≥10% Weight Loss at Month 6 | Month 6
  Percentage of participants with ≥10% weight loss at month 6.
Mean Percent Change of Weight from Baseline | Baseline, Month 6 and Baseline, Month 12
  Mean percent change of weight from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (55):
- United States (53):
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Avondale, Avondale, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Chandler, Chandler, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Flagstaff, Flagstaff, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Gilbert, Gilbert, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Glendale, Glendale, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Mesa, Mesa, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Phoenix PV, Phoenix, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Sun City, Sun City, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Tucson, Tucson, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Tucson Southeast, Tucson, Arizona
  - Medvin Clinical Research - Apple Valley, Apple Valley, California
  - Medvin Clinical Research - Covina, Covina, California
  - Newport Huntington Medical Group, Huntington Beach, California
  - Purushotham & Akther Kotha MD, Inc, La Mesa, California
  - Medvin Clinical Research - Riverside, Riverside, California
  - Rheumatology Center of San Diego, San Diego, California
  - Providence Saint John's Medical Foundation, Santa Monica, California
  - Medvin Clinical Research - Temecula, Temecula, California
  - Medvin Clinical Research - Tujunga, Tujunga, California
  - Medvin Clinical Research - Whittier, Whittier, California
  - Vida Clinical Research, Kissimmee, Florida
  - Life Clinical Trials, Margate, Florida
  - CZ Rheumatology, Miami Beach, Florida
  - Vitalia Medical Research, Palm Beach Gardens, Florida
  - International Center for Research, Tampa, Florida
  - Atlanta Research Center for Rheumatology, Marietta, Georgia
  - Satilla Rheumatology & Internal Medicine, Waycross, Georgia
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Greater Chicago Specialty Physicians, Schaumburg, Illinois
  - Arnold Arthritis & Rheumatology, Skokie, Illinois
  - Willow Rheumatology and Wellness PLLC, Willowbrook, Illinois
  - Lake Cumberland Rheumatology, New Albany, Indiana
  - Accurate Clinical Research, Inc, Lake Charles, Louisiana
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - Logan Health Rheumatology, Kalispell, Montana
  - University of Rochester Medical Center, Rochester, New York
  - Onsite Clinical Solutions, LLC - Brenner Ave, Salisbury, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Essential Medical Research, Tulsa, Oklahoma
  - West Tennessee Research Institute, Jackson, Tennessee
  - AARA Clinical Research - Murfreesboro Medical Clinic, Murfreesboro, Tennessee
  - Precision Comprehensive Clinical Research Solutions - Colleyville, Colleyville, Texas
  - AARA Clinical Research - Lone Star Arthritis and Rheumatology Associates - Fort Worth, Fort Worth, Texas
  - Accurate Clinical Research, Inc, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - AARA Clinical Research - Lone Star Arthritis and Rheumatology Associates - Irving, Irving, Texas
  - Biopharma Informatic, LLC, Katy, Texas
  - Advanced Rheumatology of Houston - Woodlands, The Woodlands, Texas
  - DM Clinical Research - TRA, Tomball, Texas
  - Seattle Rheumatology Associates PLLC, Seattle, Washington
  - Arthritis Northwest, PLLC, Spokane Valley, Washington
- Puerto Rico (2):
  - Reuviva Research Center, Guaynabo
  - CMRC Headlands, LLC, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Plan Description: Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/580115